CLINICAL TRIAL: NCT02002650
Title: Routine Rectal Indomethacin Given Before Procedure Reduced Overall Pancreatitis in Patients Undergoing Endoscopic Retrograde Cholangiopancreatography (ERCP): A Multi-center, Single-blinded, Randomized Controlled Trial
Brief Title: Rectal Indomethacin to Prevent Post-ERCP Pancreatitis
Acronym: Indomethacin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Yanglin Pan, Associated professor, Air Force Military Medical University, China
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 20131106-7; 20131106-7 (Other: Ethics committee of Xijing Hospital)
Record Dates: First submitted 2013-12-01; First posted 2013-12-06 (Estimated); Results first posted 2016-05-27 (Estimated); Last update posted 2016-06-29 (Estimated); Status verified 2016-05

CONDITIONS: Post-ERCP Acute Pancreatitis
Keywords: Indomethacin, pancreatitis, ERCP
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pre-ERCP group (Experimental): Pre-ERCP rectal Indomethacin in all patients.
  Interventions: Drug: Pre-ERCP rectal Indomethacin
- Post-ERCP group (Active Comparator): Post-ERCP rectal Indomethacin in high-risk patients.
  Interventions: Drug: Post-operational Rectal Indomethacin

INTERVENTIONS:
Drug: Pre-ERCP rectal Indomethacin — Rectal Indomethacin was administrated within 30min before ERCP in all patients.
  Arms: Pre-ERCP group
Drug: Post-operational Rectal Indomethacin — Rectal Indomethacin was administrated immediately after ERCP in high-risk patients, while average risk patients did not.
  Arms: Post-ERCP group

SUMMARY:
Acute pancreatitis is the most common and feared complication of ERCP, occurring after 1% to 30% of procedures. Since 2012, a multicenter RCT was published in NEJM, indomethacin use in high risk patients was considered a "standard" method to prevent PEP. However, the risk factors of PEP is not fully clear. Rectal indomethacin before ERCP for all patients, not just for selected high-risk patients, may preventing PEP maximum. The purpose of this study is to determine whether routine using of rectal indomethacin is more effective than the conditional strategy.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing diagnostic or therapeutic ERCP.

Exclusion Criteria:

* Unwillingness or inability to consent for the study;
* Age < 18 years old;
* Intrauterine pregnancy;
* Breastfeeding mother;
* Standard contraindications to ERCP;
* Allergy to NSAIDs;
* Received NSAIDs in prior 7 days;
* Renal failure (Cr >1.4mg/dl=120umol/l);
* Active or recurrent (within 4 weeks) gastrointestinal hemorrhage;
* Acute pancreatitis within 72 hours;
* Known pancreatic head mass;
* Subject with prior biliary sphincterotomy now scheduled for repeat biliary therapy without anticipated pancreatogram;
* ERCP for biliary stent removal or exchange without anticipated pancreatogram;
* Known active cardiovascular or cerebrovascular disease.
* Presence of coagulopathy before the procedure or received anticoagulation therapy within three days before the procedure;

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2600 (Actual)
Dates: Start 2013-12; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yanglin Pan, M.D., Study Director — Xijing Hospital of Digestive Diseases.The Fourth Military Medical University
Locations (6):
- China (6):
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - General Hospital of NingXia Medical University, Yinchuan, Ningxia
  - Xijing Hospital of Digestive Diseases, Xi'an, Shaanxi
  - No. 451 Hospital, Xi'an, Shaanxi
  - The First Affiliated Hospital Of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Urumqi General Hospital of Lanzhou Military Region, Ürümqi, Xinjiang

REFERENCES:
- [Result] Ding X, Chen M, Huang S, Zhang S, Zou X. Nonsteroidal anti-inflammatory drugs for prevention of post-ERCP pancreatitis: a meta-analysis. Gastrointest Endosc. 2012 Dec;76(6):1152-9. doi: 10.1016/j.gie.2012.08.021. PMID 23164513
- [Result] Elmunzer BJ, Scheiman JM, Lehman GA, Chak A, Mosler P, Higgins PD, Hayward RA, Romagnuolo J, Elta GH, Sherman S, Waljee AK, Repaka A, Atkinson MR, Cote GA, Kwon RS, McHenry L, Piraka CR, Wamsteker EJ, Watkins JL, Korsnes SJ, Schmidt SE, Turner SM, Nicholson S, Fogel EL; U.S. Cooperative for Outcomes Research in Endoscopy (USCORE). A randomized trial of rectal indomethacin to prevent post-ERCP pancreatitis. N Engl J Med. 2012 Apr 12;366(15):1414-22. doi: 10.1056/NEJMoa1111103. PMID 22494121
- [Derived] Luo H, Zhao L, Leung J, Zhang R, Liu Z, Wang X, Wang B, Nie Z, Lei T, Li X, Zhou W, Zhang L, Wang Q, Li M, Zhou Y, Liu Q, Sun H, Wang Z, Liang S, Guo X, Tao Q, Wu K, Pan Y, Guo X, Fan D. Routine pre-procedural rectal indometacin versus selective post-procedural rectal indometacin to prevent pancreatitis in patients undergoing endoscopic retrograde cholangiopancreatography: a multicentre, single-blinded, randomised controlled trial. Lancet. 2016 Jun 4;387(10035):2293-2301. doi: 10.1016/S0140-6736(16)30310-5. Epub 2016 Apr 28. PMID 27133971

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From Dec 15, 2013 to Sep 21, 2015, 5325 consecutive patients undergoing ERCP in six centers in China were considered for the study.
Pre-assignment Details: After screening, 2725 patients were excluded: 193 did not meet inclusion criteria, 2304 met exclusion criteria and 228 patients declined to participate.
Groups:
- Post-ERCP Group: Post-ERCP rectal Indomethacin in high-risk patients.
  Post-ERCP Rectal Indomethacin: Rectal Indomethacin was administrated immediately after ERCP just in high-risk patients, while average risk patients did not.
Period: Overall Study
Arm/Group | Pre-ERCP Group | Post-ERCP Group
Started | 1297 | 1303
Completed | 1297 | 1303
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Pre-ERCP Group: Pre-ERCP rectal Indomethacin in all patients.
  Pre-operational rectal Indomethacin: Rectal Indomethacin was administrated within 30min before ERCP in all patients.
- Total: Total of all reporting groups
Arm/Group | Pre-ERCP Group | Post-ERCP Group | Total
Number analyzed (Participants) | 1297 | 1303 | 2600
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 62 [50 to 72] | 63 [50 to 74] | 62 [50 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 688 | 693 | 1381
  Male | 609 | 610 | 1219
High-risk patients [Number; unit: participants] — met at least one of the major criteria - clinical suspicion of sphincter of Oddi dysfunction, a history of PEP, pancreatic sphincterotomy, precut sphincterotomy, ≥8 cannulation attempts, pneumatic dilatation of an intact biliary sphincter, or ampullectomy.
  or met two or more of the minor criteria - age<50 and female gender, a history of recurrent pancreatitis (≥2 episodes), ≥3 injections of contrast into the pancreatic duct with ≥1 injection to the tail of the pancreas, opacification of pancreatic acini, or brush cytology performed on the pancreatic duct.
  participants | 305 | 281 | 586

OUTCOME MEASURES:

1. Primary Outcome: Post-ERCP Pancreatitis
Description: Subjects were diagnosed with post-ERCP pancreatitis if they experienced new upper abdominal pain, serum amylase elevation at least three times the upper limit of normal 24 hours after the procedure, and hospitalization prolonged at least two nights.
Time Frame: 30 days
Measure: Number; unit: participants
Arm/Group | Pre-ERCP Group | Post-ERCP Group
Number analyzed (Participants) | 1297 | 1303
participants | 47 | 100

2. Secondary Outcome: Moderate-to-severe Pancreatitis
Description: Moderate pancreatitis requiring hospitalization of 4-10 days. Severe pancreatitis requiring hospitalization for more than 10 days, or hemorrhagic pancreatitis, phlegmon or pseudocyst, or intervention (percutaneous drainage or surgery).
Time Frame: 30 days
Measure: Number; unit: participants
Groups:
- Post-ERCP Group: Post-ERCP rectal Indomethacin for high-risk patients.
  Post-ERCP Rectal Indomethacin: Rectal Indomethacin was administrated immediately after ERCP just for high-risk patients.
Arm/Group | Pre-ERCP Group | Post-ERCP Group
Number analyzed (Participants) | 1297 | 1303
participants | 11 | 23

ADVERSE EVENTS:
Time Frame: 30 days
Description: Adverse events related to ERCP or indomethacin include bleeding, perforation, biliary infection, cardiovascular or renal adverse events and other adverse events.
Arm/Group | Pre-ERCP Group | Post-ERCP Group
Serious Adverse Events (participants affected / at risk) | 15/1297 | 15/1303
Other Adverse Events (participants affected / at risk) | 26/1297 | 33/1303
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pre-ERCP Group (N=1297) | Post-ERCP Group (N=1303)
Moderate to severe bleeding (Gastrointestinal disorders) | 8 (8) | 6 (6) — Moderate to severe bleeding was defined as clinically significant bleeding with hemoglobin level drop ≥3g with the need for transfusion, angiographic intervention or surgery.
Moderate to severe biliary infection (Infections and infestations) | 7 (7) | 9 (9) — Febrile or septic illness requiring >3 d of hospital treatment or need endoscopic or percutaneous intervention. Septic shock or surgery.
OTHER ADVERSE EVENTS (reported when occurring in more than 0.01% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pre-ERCP Group (N=1297) | Post-ERCP Group (N=1303)
Mild bleeding (Gastrointestinal disorders) | 5 (5) | 4 (4) — Clinical evidence of bleeding (ie, not just endoscopic); Hb level drop <3 g; no need for transfusion.
Mild biliary infection (Infections and infestations) | 15 (15) | 24 (24) — Mild biliary infection was defined as a temperature of more than 38°C for 24-48 h after the procedure, thought to have a biliary cause (colicky pain and cholestasis/jaundice) without evidence of other concomitant infections.
Mild perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) — Possible, or only very slight leak of fluid or contrast dye; treatable by fluids and suction for ≤3d
Pulmonary infection (Infections and infestations) | 2 (2) | 5 (5)
Incomplete bowel obstruction (Gastrointestinal disorders) | 3 (3) | 0 (0)

LIMITATIONS AND CAVEATS:
Firstly, patients could not be blinded to the treatment assignment. Secondly, it remains unclear if patients with prior EST will benefit from rectal indomethacin. Thirdly, the findings need to be validated in different clinical settings.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No